CLINICAL TRIAL: NCT03737461
Title: A Phase 2/3 Prospective, Multicentre Randomized, Double-blind Trial, Comparing Intra-discal Allogeneic Adult BM-MSC Therapy and Sham-treated Controls in Subjects With Chronic LBP Due to Lumbar DDD Unresponsive to Conventional Therapy
Brief Title: Efficacy of Intradiscal Injection of BM-MSC in Subjects With Chronic Low Back Pain (LBP) Due to Lumbar Degenerative Disc Disease (DDD) Unresponsive
Acronym: RESPINE
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Interdisziplinäres Zentrum Klinische Studien (IZKS) (Unknown); European Clinical Research Infrastructure Network (Other); Département de l'information médicale, CHU de Montpellier (Unknown); Centre National de la Recherche Scientifique, France (Other); Université Montpellier (Other); Univercell-Biosolutions S.A.S (Unknown); National University of Ireland, Galway, Ireland (Other); University of Valladolid (Other); Citospin (Industry); Rennes University Hospital (Other); APHP (Other); Campus Bio-Medico University (Other); BG Klinikum Bergmannstrost, Halle, Germany (Unknown); Nantes University Hospital (Other); Institut de Terapia Regenerativa Tissular (Other); University of Navarra (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RECHMPL17_0206; 2017-002092-25 (EudraCT Number)
Record Dates: First submitted 2018-06-19; First posted 2018-11-09 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Recurrent Low Back Pain; Degenerative Disc Disease (DDD)
Keywords: BM-MSCs; Low back pain; Lumbar degenerative disc disease (DDD)
MeSH Terms: conditions — Low Back Pain; Intervertebral Disc Degeneration | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Allogenic BM-MSCs Injection (Experimental): Injection of a dose of 20.106 allogenic BM-MSCs via imaging control into the disk affected by DDD where they are expected to exert their therapeutic effects.
  Interventions: Drug: Allogenic BM-MSCs Injection
- Sham Procedure (Sham Comparator): anesthetic infiltration with 2 ml of 1% xylocaine in the paravertebral muscles close to the affected segment
  Interventions: Other: Sham Procedure

INTERVENTIONS:
Drug: Allogenic BM-MSCs Injection — Cell dose will be 20±5 million cells suspended in 2 ml of HypoThermosol isotonic transport solution
  Arms: Allogenic BM-MSCs Injection
Other: Sham Procedure — sham-maneuver as in the cell-treated patients are added, consisting in anesthetic infiltration with 2 ml of 1% xylocaine in the paravertebral muscles close to the affected segment.
  Other Names: Injection of 2 mL of 1% xylocaine
  Arms: Sham Procedure

SUMMARY:
This will be a multicenter, prospective, double blind, randomized phase 2/3 trial comparing culture-expanded allogeneic adult BM-MSCs with sham-treated controls.

This trial will evaluate the efficacy of intradiscal injection of BM-MSCs in chronic low back pain due to lumbar degenerative disc disease (DDD) unresponsive to conventional therapy .

Visual analog scale (VAS) and functional status (by Oswestry Disability Index - ODI) will be evaluated 12 months after treatment, defining responders in case of improvement of VAS for pain of at least 20% and 20 mm between baseline and month 12, or improvement of ODI of 20% between baseline and month 12.

DETAILED DESCRIPTION:
Degenerative disc disease (DDD) presents a large, unmet medical need. One of the most important public health problems, it affects 70 million Europeans, accounts for 42% of patients with chronic low back pain and costs over $100 billion each year in the European Union. DDD results in a disabling loss of mechanical function. Today, no efficient therapy is available. The disease results from degeneration of cartilage discs with loss of the collagen matrix and nucleus pulposus chondrocyte. Chronic cases often receive surgery, which may lead to biomechanical problems and accelerated degeneration of adjacent segments. Our consortium partners have developed and studied stem cell-based, regenerative therapies with encouraging results in phase 1 and 2 trials. Patients exhibited rapid and progressive improvement of functional and pain indexes by 50% within 6 months and by 65% to 78% after 1 year with no side effects. In addition, MRI T2 relaxation measurements demonstrated a significant improvement of cartilage signal. To develop the world's first effective treatment of DDD, RESPINE aims to assess, via a randomized, controlled, phase 3 clinical trial including 112 patients with DDD, the efficacy of an allogenic intervertebral mesenchymal stem cell (MSC)-based therapy. This innovative therapy aims to rapidly (within 3 months) and durably (at least 24 months) reduce pain and disability. In addition, the consortium aims to provide new knowledge on immune response & safety associated with allogeneic BM-MSC intradiscal injection.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 60 years.
* Symptomatic chronic low back pain unresponsive to conservative therapy (including physical therapy performed during at least 1 month before inclusion and pain medication with level 2 analgesics in failure or intolerant to level during at least 1 month) for at least 3 months.
* DDD assessed by (Pfirrmann's score modified Griffith et al) grade 4 to 7 at one level. If second level, it should be adjacent (Pfirrmann's score 1-4 maximum)
* Low back Pain baseline > 40 mm on VAS (0-100).
* NSAID washout of at least 2 days before screening
* Painkillers washout of at least 24 hours before screening

Exclusion Criteria:

* Congenital or acquired diseases leading to spine deformations that may upset cell application (hyperlordosis, scoliosis, isthmus lesion, sacralization and hemisacralization).
* Symptomatic posterior lumbo-articular osteoarthritis or predominant facet syndrome on Xray or MRI (osteophyte and facet hypertrophy).
* Prior to the screening visit, has received:
* Oral corticosteroid therapy within the previous 3 months, OR
* Intramuscular, intravenous or epidural corticosteroid therapy within the previous 3 months
* Spinal segmental instability (defined by lumbar dynamic X-Ray in extension/flexion with antero-post translation > 3 mm and/or angular mobility > 15°).
* Spinal canal stenosis (Schizas score > B).
* History of spinal infection.
* Lumbar disc herniation with non truncated sciatica or cruralgia, as well as lumbar cysts and radiculopathy
* Previous discal puncture or previous spine surgery.
* DDD on 3 levels, or DDD on 2 levels but not adjacent, or DDD with modic 2 or 3 phases
* Patients not eligible to the intravertebral disc surgery
* Patients who have the risk to undergo a surgery in the next 6 months
* Obesity with body mass index (BMI in Kg/size in m2) greater than 35 (obesity grade II).
* Participation in another clinical trial or treatment with another investigational product within 30 days prior to inclusion in the study.
* Abnormal blood tests: hepatic (alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) >1.5 × upper limit of normal (ULN)), renal, pancreatic or biliary disease, blood coagulation disorders, anemia or platelet count of <100 × 109/
* Significant medical problems, such as uncontrolled hypertension, symptomatic heart failure; or any other clinically relevant condition or current medication that in the opinion of the investigator contra-indicates the use of any of the study or rescue medications.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 113 (Actual)
Dates: Start 2019-02-18 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2026-03-08 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Pain Clinical response at 12 months | baseline to month 12
  The clinical response is defined as the Pain relief measure with Visual Analogue Scale (VAS) of at least 20 mm decrease on VAS scale between baseline and month 12.
Change from Baseline Oswestry Disability Index (ODI) measure at 12 months | baseline to month 12
  at least 20% improvement of functional index ODI at month 12 compared to baseline.

SECONDARY OUTCOMES:
Measure disability and quality of life evolution of the patient | Baseline, 3,6,12 and 24 months
  Assessed by Short Form-36 Health Survey (SF-36) :
  The eight sections are vitality, physical functioning, bodily pain, general health, perceptions, physical role functioning, emotional role functioning, social role functioning and mental health A score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Disability and quality of life evolution | baseline, 3,6,12 and 24 months
  global assessment by the patient and the physician. Overall pain intensity in the lumbar spine (1 = none, 2 = mild, 3 = moderate, 4 = severe, 5 = extreme); patient's global assessment of disease activity (1 = very good, 2 = good, 3 = fair, 4 = poor, 5 = very poor); physician's global assessment of disease activity (1 = very good, 2 = good, 3 = fair, 4 = poor, 5 = very poor) will be performed at 0, 3, 6, 12 and 24 months.
Pain killers | baseline, 1, 3,6,12 and 24 months
  assessement of consumption of painkillers medication. Rescue medication use will be recorded throughout the study duration by a diary file.
Measure of the Chronic low back pain | baseline, 1, 3,6,12 and 24 months
  assessement of pain by the Visual Analogue pain Scale (VAS) during 24 months. Min value 0 - max value 100 , where 0 represents no pain and 100 represents the worst pain imaginable.
Employment and work status | baseline, 1, 3,6,12 and 24 months
  Assessement of employment and work status. For this, patients will be assign to one of 4 categories designated as "employable" which included those who were unemployed due to pain, employed but on sick leave, laid off, or working. The other categories include retired, disabled, and elderly at least 60 years of age, eligible for social security.
Structural assessment | baseline, 1, 3,6,12 and 24 months
  Evolution of affected disc(s) by quantitative Magnetic Resonance Imaging (MRI) density measurements in T2 and T1spin/echo and T1rho weighted images performed at 0, 6 12 and 24 months used as an indication of disc fluid and glycosaminoglycan (GAG) content. The "quality" of the patient's lumbar disc will be monitored non invasively using T2-weighted MRI sagittal images (Orozco et al., 2011) and, in T1spin/echo MRI. Lumbar disc grading will be performed in the sagittal T2 weighted images by two physicians independently who were experienced in MRI of the spine. They will review each intervertebral disc from L1-2 to L5-S1 by the modified Pfirrmann criteria. The modified Pfirrmann grading system assesses degenerated intervertebral discs by MRI for the asymmetry in disc structure, distinction of the nucleus and the annulus, signal intensity of intervertebral discs and height of intervertebral discs and assigns grade 1 to 8 for disc degeneration (Table by Griffin et al. Spine 2007).
Evaluation of cost | 24 months
  We will compare the medical and non-medical costs between the two groups of patient. Costs will be identified for a one-year time horizon.
  For this purpose, resource use in each arm will be collected in physical units in the electronic Case Report Form (eCRF) at each clinical centre as follows:
  * Acute care medical hospitalisations related to DDD
  * Acute care surgical hospitalisations related to DDD
  * Rehabilitation hospitalisations related to DDD
  * Analgesics
  * Work disruption Resource use will be valued using production costs specific to each country or to the country having included the highest number of patients, depending on the number of patients actually included in each clinical centre.
Immune response / Analytical control | baseline, 1, and 6 months
  The assessment of the biological effect of allogeneic MSC on recipient immune response will be studied by multiparametric flow-cytometry as well as monitoring of anti HLA-I (human leukocyte antigen I) antibodies response.
reporting of Serious Adverse Events (SAE) | baseline, 1, 3,6,12 and 24 months
  Define the safety outcomes of the clinical trial with the record of SAE

CONTACTS AND LOCATIONS:
Overall Officials: Christian CJ JORGENSEN, PhD, Principal Investigator — Montpellier University Hospital
Locations (9):
- France (4):
  - UH Montpellier, Montpellier
  - CHU de Nantes, Nantes
  - CHU Saint Antoine, Paris
  - APHP Cochin, Paris
- BG Klinikum Bergmannstrost, Halle, Germany
- Campus Bio-Medico University of Rome, Roma, Italy
- Spain (3):
  - Institut de Teràpia Regenerativa Tissular, Barcelona
  - Clínica Universidad de Navarra, Pamplona
  - Hospital Sagrado Corazón Valladolid, Valladolid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pers YM, Soler-Rich R, Vadala G, Ferreira R, Duflos C, Picot MC, Herman F, Broussous S, Sanchez A, Noriega D, Ardura F, Alberca Zaballos M, Garcia V, Gordillo Cano V, Gonzalez-Vallinas M, Denaro V, Russo F, Guicheux J, Vilanova J, Orozco L, Meisel HJ, Alfonso M, Rannou F, Maugars Y, Berenbaum F, Barry FP, Tarte K, Louis-Plence P, Ferreira-Dos-Santos G, Garcia-Sancho J, Jorgensen C; RESPINE consortium. Allogenic bone marrow-derived mesenchymal stromal cell-based therapy for patients with chronic low back pain: a prospective, multicentre, randomised placebo controlled trial (RESPINE study). Ann Rheum Dis. 2024 Oct 21;83(11):1572-1583. doi: 10.1136/ard-2024-225771. PMID 39393844